CLINICAL TRIAL: NCT05947539
Title: Improving HIV Care Engagement Among Ugandan Adolescent Girls and Young Women Through Reductions in Male Partner Alcohol Use and Intimate Partner Violence Risk: The Kisoboka Mukwano Intervention
Brief Title: Improving HIV Care Engagement Among Ugandan Adolescent Girls and Young Women: The Kisoboka Mukwano Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); San Diego State University (Other); Makerere University (Other); University of California, San Diego (Other); Reach the Youth Uganda (Other)
Responsible Party: Principal Investigator, Ijeoma Ogbonnaya, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R34AA030489 (NIH); R34AA030489 (NIH)
Record Dates: First submitted 2023-03-22; First posted 2023-07-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-08

CONDITIONS: HIV-infection/Aids; Intimate Partner Violence; Domestic Violence; Alcohol Use Disorder
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcoholism | interventions — Methods; Mass Screening; Referral and Consultation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kisoboka Mukwano Intervention (treatment) (Experimental): A brief couples-based intervention using motivational interviewing, peer navigation, and behavioral economic approaches to target intimate partner violence, alcohol use, and HIV care engagement.
  Interventions: Behavioral: Kisoboka Mukwano ("It is possible, my love!") Intervention
- Screening & Referral (control) (Active Comparator): Brief feedback on intimate partner violence and alcohol use (males), referrals for these conditions, and briefly discuss the importance of HIV care engagement and adherence.
  Interventions: Behavioral: Screening and Referral

INTERVENTIONS:
Behavioral: Kisoboka Mukwano ("It is possible, my love!") Intervention — The intervention consists of 5 bi-weekly sessions each lasting 60 to 90 minutes. It uses motivational interviewing, peer navigation, and behavioral economics to promote strategies for economic strengthening, reductions in male partner alcohol use, coping with relationship conflict and stress, changing norms that reduce intimate partner violence and support engagement in HIV care and antiretroviral therapy (ART) adherence among adolescent girls and young women living with HIV, and, thereby, enhances future sustained viral suppression and benefits of treatment as prevention.
  Arms: Kisoboka Mukwano Intervention (treatment)
Behavioral: Screening and Referral — Intimate partner violence screening, alcohol screening, and referral
  Arms: Screening & Referral (control)

SUMMARY:
This study will develop and pilot test a couples-based intervention to help adolescent girls and young women living with HIV (WLHIV (15-24 years) living in Uganda access HIV care and improve the outcomes of their HIV treatment by targeting male partner alcohol use to reduce IPV risk.

DETAILED DESCRIPTION:
In Uganda, adolescent girls and young women (AGYW) are disproportionately affected by HIV and have poor viral suppression rates, increasing their risk of onward transmission. Intimate partner violence (IPV) is a major barrier to mitigating the impact of HIV among AGYW. AGYW living with HIV (AGYWLHIV) in sub-Saharan Africa (SSA) who have experienced IPV have worse medication adherence, viral suppression, and care engagement than those without IPV. Further, male partner alcohol use directly and indirectly increases IPV risk among AGYW in SSA. Thus, an intervention with components that address heavy alcohol use among male partners could decrease AGYW's IPV risk, especially in Uganda, which has the highest alcohol use per capita in SSA. Couples- based interventions have effectively reduced male partner alcohol use, relationship conflict IPV, and improved viral suppression and HIV care engagement; yet, none have been tailored to AGYWLHIV in SSA. The investigators propose to develop and pilot a couples-based intervention that focuses on improving HIV care engagement and ART adherence among AGYWLHIV by reducing heavy alcohol use among male partners and couple IPV risk. Additionally, the investigators will explore the intervention's effects on AGYW viral load for the additional key benefit of treatment as prevention. The study aims are to: 1) Adapt the behavioral components of a brief Motivational Interviewing (MI)-based alcohol intervention to create the proposed Kisoboka Mukwano ("It is possible, my love!") intervention. The intervention will promote strategies for reductions in male partner alcohol use, coping with relationship conflict and stress, changing norms that reduce IPV and support engagement in HIV care and ART adherence among AGYWLHIV, and, thereby, enhance future sustained viral suppression and benefits of treatment as prevention. The intervention will be adapted and tailored to be delivered with heterosexual couples, involve peer navigators, address IPV, and be developmentally appropriate for AGYWLHIV in Uganda. The investigators will develop and refine the intervention in collaboration with an intervention steering committee through: qualitative research with married/cohabiting AGYWLHIV, married/cohabiting men, and key informants and an initial pilot test with 6 couples. 2) The investigators will assess safety, acceptability, feasibility, and preliminary estimates of the potential for the intervention, as compared to the control group, to improve HIV, alcohol, and IPV outcomes. The investigators will examine preliminary effects on AGYW HIV care engagement, AGYW ART adherence, heavy alcohol use among male partners, and couple IPV risk and explore effects on AGYW viral load as well as intermediate outcomes related to intervention components. The investigators will assess these outcomes at baseline and then at 3- and 6-month follow-up. Study findings will be used to guide a subsequent R01 proposal to test the intervention in a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria

Adolescent girls and young women (AGYW)/Female:

* aged 18-24 or self-reported as emancipated minors aged 15-17,
* HIV+
* meets one or more of the following non-engagement criteria: not currently enrolled in an HIV clinic (e.g., never enrolled, dropped out); not currently taking ART; missed 1 or more scheduled HIV care appointments requiring physical presence (e.g., viral load [VL] testing) in the last 12 months; < 90% ART adherence in the last 2 weeks; most recent VL>1000 or expected recent VL test results absent in clinic records despite initiating ART >6 months ago
* self-report a history of at least one incident of IPV (physical, sexual, and/or emotional) and/or controlling behavior ever perpetrated by their current male partner
* agree to let research staff contact their male partner.

Male Partners of AGYW/Male:

* aged 18+ years or emancipated minors
* report consuming ≥ 6 drinks per occasion at least once or more in the prior 30 days or scores 4 or more on the AUDIT (Alcohol Use Disorders Identification Test)-C

Couples (each partner (male and female) must independently report):

* married or living together as if married for ≥6 months
* planning to stay together for at least another 2 months (intervention period)
* lived in the Wakiso District area ≥3 months
* not planning to move from the area within the next 6 months
* respond similarly (not exact but close) to questions on the study-developed Couple Verification Screening

Exclusion Criteria

AGYW (female):

* reporting any severe physical IPV experienced in prior 3 months.

Couples (male and female):

* do not speak Luganda or English
* do not feel they cannot safely participate in the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
change from baseline in antiretroviral therapy (ART) adherence biomarker (females and HIV+ male partners) | 3 and 6 month follow up
  presence of Tenofoivir Disoproxil Fumarate (TDF) detected in urine
change from baseline in self-reported antiretroviral therapy (ART) adherence (females and HIV+ male partners) | 3 and 6 month follow up
  Self- report of missed ART using the AIDS Clinical Trials Group Adherence (AACTG) measures
change from baseline in HIV care engagement (females and HIV+ male partners) | 3 months, 6 months
  HIV clinic visit adherence
change from baseline in phosphatidylethanol (PEth) (male partners) | 6 months
  alcohol biomarker (PEth) levels
change from baseline in heavy drinking (male partners) | 3 months, 6 months
  assessed with the Alcohol Use Disorders Identification Test (AUDIT-C)
Intimate partner violence (IPV) occurence (males and females) | 6 months
  Any incident of IPV perpetration and victimization: physical, sexual, verbal/emotional, intimidation and/or controlling behavior measured using the World Health Organization (WHO) Instrument/ Demographic and Health Data (DHS) Domestic Violence Modules.

SECONDARY OUTCOMES:
Fear of intimate partner violence (males and females) | 6 month follow up
  Rating of how often one is afraid of their current spouse/partner measured using the WHO Instrument/ DHS Domestic Violence Modules.

OTHER OUTCOMES:
change from baseline in HIV viral load (females and HIV+ males) | 6 months
  (1) Biomarker testing using blood (females) and (2) clinic records (males).
change from baseline in PrEP adherence (male partners taking PrEP) | 3 and 6 month follow up
  self- report of missed PrEP using an adapted version of the AIDS Clinical Trials Group Adherence (AACTG) measures
PrEP uptake | through 6 month follow-up
  Initiation of PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Ijeoma Nwabuzor Ogbonnaya, PhD, Principal Investigator — Arizona State University; Susan M Kiene, PhD, Principal Investigator — San Diego State University
Locations (1):
- Makerere Univerisity School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) that underlie the 6-month clinical trial, excluding qualitative data and data collected for formative research.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Two years after the grant end date specified on the first Notice of Award (08-31-2025). Any subject-level data and the associated analyzed data used in a journal publication will be shared at the time of publication, even if the publication occurs before the two-year automatic share date.
Access Criteria: Access to data for research purposes will be provided through the National Institute of Mental Health (NIMH) Data Archive (NDA) Data Access Committee (DAC). Investigators and institutions seeking data from NDA will be expected to meet data security measures and will be asked to submit a Data Use Certification, which is cosigned by the investigator and the designated Institutional Official(s) at the NIH-recognized sponsoring institution with a current Federal Wide Assurance (FWA).
URL: https://nda.nih.gov/nda/standard-operating-procedures.html#sop4a

REFERENCES:
- [Derived] Nwabuzor Ogbonnaya I, Nakigudde J, Naigino R, Stockman JK, Chung Y, Nantongo M, Marsiglia FF, Hahn JA, Wechsberg WM, Mwebembezi A, Wanyenze RK, Kiene SM. Protocol for the Kisoboka Mukwano pilot randomized controlled trial in Uganda: A couples-based intervention to reduce intimate partner violence and alcohol use among adolescent girls and young women living with HIV and their male partners. Contemp Clin Trials. 2025 Dec;159:108136. doi: 10.1016/j.cct.2025.108136. Epub 2025 Nov 7. PMID 41207472

DOCUMENTS (1):
  • Informed Consent Form (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT05947539/ICF_000.pdf